CLINICAL TRIAL: NCT01442883
Title: Understanding the Mechanisms of Progressive Decrease in Blood Pressure After Renal Nerve Ablation
Brief Title: Renal Nerve Ablation in Chronic Kidney Disease Patients
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: RNA-CKD3-5
Record Dates: First submitted 2011-09-22; First posted 2011-09-29 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Hypertension; Chronic Kidney Disease
Keywords: Treatment Resistant
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- treatment resistant hypertensives with CKD 3-5
  Interventions: Device: Simplicity Catheter

INTERVENTIONS:
Device: Simplicity Catheter — percutaneous selective renal sympathetic nerve ablation with the use of the Simplicity Catheter system

SUMMARY:
In patients with treatment resistent hypertension renal nerve ablation emerged as an effective interventional approach of treating hypertensive disease with a progressively increasing fall in blood pressure. Decreased activity of the sympathetic nervous system is one of the major underlying pathogenetic mechanism of the fall in blood pressure but the precise mechanisms that causes the fall in blood pressure in the short-term and, in particular, long-term remains elusive. The objective of the study is to understand the pathogenetic mechanisms of renal denervation beyond the reduced activity of the sympathetic nervous system. In 100 hypertensive patients most advanced technology will be applied, before and repeatedly after renal denervation, throughout the follow-up period of 1 year. Systemic activity of the renin angiotensin aldosterone system, renal perfusion (by MRI spin labelling technique), local activity of the renin angiotensin system in the kidney (urinary angiotensinogen concentrations), sodium excretion and total sodium content (23 Na-MRI technique) and vascular remodelling of small (retinal arterioles 50 - 150 µm) and large arteries (carotid - femoral pulse wave velocity and augmentation index, both measured over 24 hours) will be assessed. Identification of the pathogenetic mechanisms involved in the fall in blood pressure after renal denervation may help to identify those hypertensive patients that profit most from renal nerve ablation in terms of blood pressure reduction.

The investigators propose the following hypotheses why a progressive decrease in blood pressure happens, in addition to the decreased activity of the central nervous system, after renal nerve ablation:

Short term effects:

A)Preservation of renal function and perfusion B)Reduction of local RAS activity in the kidney C)Exaggerated sodium excretion immediately after renal nerve ablation

Long term effects:

D)Decrease of total sodium content after 6 and 12 months. E)Improvement of vascular wall properties after 6 and 12 months

DETAILED DESCRIPTION:
In patients with treatment resistent hypertension renal nerve ablation emerged as an effective interventional approach of treating hypertensive disease with a progressively increasing fall in blood pressure. Decreased activity of the sympathetic nervous system is one of the major underlying pathogenetic mechanism of the fall in blood pressure but the precise mechanisms that causes the fall in blood pressure in the short-term and, in particular, long-term remains elusive. The objective of the study is to understand the pathogenetic mechanisms of renal denervation beyond the reduced activity of the sympathetic nervous system. In 100 hypertensive patients most advanced technology will be applied, before and repeatedly after renal denervation, throughout the follow-up period of 1 year. Systemic activity of the renin angiotensin aldosterone system, renal perfusion (by MRI spin labelling technique), local activity of the renin angiotensin system in the kidney (urinary angiotensinogen concentrations), sodium excretion and total sodium content (23 Na-MRI technique) and vascular remodelling of small (retinal arterioles 50 - 150 µm) and large arteries (carotid - femoral pulse wave velocity and augmentation index, both measured over 24 hours) will be assessed. Identification of the pathogenetic mechanisms involved in the fall in blood pressure after renal denervation may help to identify those hypertensive patients that profit most from renal nerve ablation in terms of blood pressure reduction.

ELIGIBILITY:
Inclusion Criteria:

* treatment resistant hypertension
* chronic kidney disease 3 - 5
* male of female aged over 18 years
* written informed consent
* agreement to attend all study visits as planned in the protocol

Exclusion Criteria:

* any contraindications for MRI
* claustrophobia
* strabismus
* severe ocular diseases
* history of epilepsia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: treatment resistant hypertensive adults with chronic kidney disease 3 - 5
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
office BP | baseline, 6 months
  Change in office blood pressure from baseline to 6 months post-renal nerve ablation
24-h ABPM | baseline, 6 months
  Change in 24 hour ambulatory blood pressure (ABPM) from baseline to 6 months post-renal nerve ablation
Magnetic resonance imaging (MRI) | baseline, 6 months
  * change in total sodium content measured by MRI from baseline to 6 months post-renal nerve ablation
  * change in renal perfusion measured by MRI spin labelling technique from baseline to 6 months post-renal nerve ablation
Albuminuria | baseline, 6 months
  Change in urinary albumin/creatinine ratio from baseline to 6 months post renal nerve ablation (spot urine)
local RAS activity | baseline, 6 months
  Change in urinary angiotensinogen concentration from the morning spot urine from baseline to 6 months post-renal nerve ablation
systemic RAS activity | baseline, 6 months
  * change in sodium, potassium and creatinine from baseline to 6 months post-renal nerve ablation
  * change in aldosterone excretion from baseline to 6 months post-renal nerve ablation
  * change in sodium / potassium ratio from baseline to 6 months post-renal nerve ablation
  * change in plasma renin activity and angiotensin II concentration at least 30 minutes of rest in a supine position and immediately after standing from baseline to 6 months post-renal nerve ablation
vascular structure and function of large and small arteries | baseline, 6 months
  * change in flow-mediated vasodilation (FMD) from baseline to 6 months post-renal nerve ablation
  * change in scanning laser Doppler flowmetry (SLDF) from baseline to 6 months post-renal nerve ablation
  * change in pulse wave analysis (PWA) from baseline to 6 months post-renal nerve ablation
  * change in pulse wave velocity from (PWV) baseline to 6 months post-renal nerve ablation
  * change in urinary albumine creatinine ratio (UACR) of the morning spot urine sample from baseline to 6 months post-renal nerve ablation

SECONDARY OUTCOMES:
BP | 1 and 12 months
  * change in office blood pressure from baseline to 1 and 12 months post-renal nerve ablation
  * change in 24 hour ambulatory blood pressure from baseline to 1 and 12 months post-renal nerve ablation
local RAS activity | 1 day and 1 months
  Change in urinary angiotensinogen concentration from the morning spot urine from baseline to 1 day and 1 months post-renal nerve ablation
systemic RAS activity | 1 day and 1 months
  * change in sodium, potassium and creatinine from baseline to 1 day and 1 months post-renal nerve ablation
  * change in albuminuria from baseline to 1 and 12 months post-renal nerve ablation
  * change in aldosterone excretion from baseline to 1 day and 1 months post-renal nerve ablation
  * change in sodium / potassium ratio from baseline to 1 day and 1 months post-renal nerve ablation
  * change in plasma renin activity and angiotensin II concentration at least 30 minutes of rest in a supine position and immediately after standing from baseline to 1 day and 1 months post-renal nerve ablation
vascular structure and function of large and small arteries | 12 months
  * change in flow-mediated vasodilation (FMD) from baseline to 12 months post-renal nerve ablation
  * change in scanning laser Doppler flowmetry (SLDF) from baseline to 12 months post-renal nerve ablation
  * change in pulse wave analysis (PWA) from baseline to 12 months post-renal nerve ablation
  * change in pulse wave velocity from (PWV) baseline to 12 months post-renal nerve ablation
  * change in urinary albumine creatinine ratio (UACR) of the morning spot urine sample from baseline to 12 months post-renal nerve ablation
MRI | 1 day, 1 and 12 months
  * change in total sodium content measured by MRI from baseline to 12 months post-renal nerve ablation
  * change in renal perfusion measured by MRI spin labelling technique from baseline to 1 day and 1 months post-renal nerve ablation

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — University of Erlangen-Nürnberg, Germany
Locations (2):
- Germany (2):
  - Clinical Research Unit, Department of Nephrology and Hypertension, University of Erlangen-Nürnberg, Erlangen
  - Joachim Weil, Lübeck

REFERENCES:
- [Background] Schmieder RE, Ott C, Schmid A, Friedrich S, Kistner I, Ditting T, Veelken R, Uder M, Toennes SW. Adherence to Antihypertensive Medication in Treatment-Resistant Hypertension Undergoing Renal Denervation. J Am Heart Assoc. 2016 Feb 12;5(2):e002343. doi: 10.1161/JAHA.115.002343. PMID 26873693
- [Background] Schmid A, Schmieder R, Lell M, Janka R, Veelken R, Schmieder RE, Uder M, Ott C. Mid-Term Vascular Safety of Renal Denervation Assessed by Follow-up MR Imaging. Cardiovasc Intervent Radiol. 2016 Mar;39(3):426-32. doi: 10.1007/s00270-015-1192-2. Epub 2015 Aug 8. PMID 26253780
- [Derived] Ott C, Mahfoud F, Schmid A, Toennes SW, Ewen S, Ditting T, Veelken R, Ukena C, Uder M, Bohm M, Schmieder RE. Renal denervation preserves renal function in patients with chronic kidney disease and resistant hypertension. J Hypertens. 2015 Jun;33(6):1261-6. doi: 10.1097/HJH.0000000000000556. PMID 25923731